CLINICAL TRIAL: NCT00880841
Title: A Single-Dose, 1-Period, 1-Treatment Pilot Study of an Investigational Capsule Formulation of 2 mg/.05 mg Buprenorphine/Naloxone Under Fasting Conditions
Brief Title: A Single-Dose Study of an Investigational Capsule Formulation of 2 mg/0.5 mg Buprenorphine/Naloxone
Status: Completed | Type: Observational
Sponsor: NanoSHIFT LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-A93-AU
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: healthy normals, phase 1; phase 1a study for healthy normals
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: phase 1a study for healthy normals
  Interventions: Drug: Buprenorphine / Naloxone

INTERVENTIONS:
Drug: Buprenorphine / Naloxone — oral formulation of buprenorphine / naloxone
  Other Names: NanoBUP

SUMMARY:
A single-dose pilot study of an investigational capsule formulation of 2 mg/.05 mg Buprenorphine/Naloxone.

NIDA Contract No. HHSN271200577414C

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breastfeeding female.
* Subject must be between 18 and 55 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects - not surgically sterile for at least 6 months or at least 2 years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal, vaginal, or injection) in use at least 3 consecutive months prior to the first dose of study medication, double barrier (condom with spermicide; diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for any outpatient visits.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, metabolic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* History or presence of allergic or adverse response to buprenorphine, naloxone, naltrexone, opioids, or any comparable or similar products.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs, such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has history of substance abuse or dependence (including alcohol, opioids, or intravenous drug abuse)
* Is a female with a positive pregnancy test result.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Has a positive urine alcohol test at screening or a positive ethanol breath test at check-in for the study period or has consumed alcohol within 48 hours prior to screening or check-in for the study period.
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C, or HIV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy normals between the ages of 18 and 55 (inclusive)
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of an investigational formulation of buprenorphine HCl/naloxone HCl 2mg/0.5mg oral capsules | pk blood draws over a 72 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Mark Leibowitz, MD, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States